CLINICAL TRIAL: NCT03712566
Title: Multi-Omic Assessment of Squamous Cell Cancers Receiving Systemic Therapy
Acronym: MASST
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: MASST-001
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Esophagus Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck; Anal Canal Squamous Cell Carcinoma; Metastatic Cancer
Keywords: Liquid Biopsy; Circulating Tumor DNA; Molecular Profiling; Immune Analysis; Epigenetics; Radiomics
MeSH Terms: conditions — Neoplasms; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected serially for DNA extraction under the LIBERATE protocol. Archived tumor samples collected for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MASST: Patients with a histological or cytological confirmed diagnosis of Squamous Cell Cancer of the Head & Neck, Esophagus or Anal Canal who have radiologically confirmed recurrent or metastatic disease and are commencing on a new treatment or either first-line platinum based chemotherapy or any line immunotherapy.

SUMMARY:
This is prospective research study which will include patients with recurrent or metastatic squamous cell carcinoma of the head and neck, esophagus and anal canal starting on first-line platinum based chemotherapy or any line of immunotherapy treatment.This study aims to characterize the dynamic changes in genomic, epigenetic, immune profiling and imaging data during treatment with systemic therapy. Patients will have archived tumor samples requested as well as blood samples collected at up to four time points to analyze these changes. Imaging data will be derived from patients' routine CT scans before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histological or cytological diagnosis of Squamous Cell Cancer of the head and neck, esophagus or anal canal who have radiologically confirmed recurrent or metastatic disease.
2. Patients must be of adequate fitness, ECOG 0-1 for systemic therapy, with either standard chemotherapy, immunotherapy or within the context of a clinical trial.
3. Patients must be commencing on a new treatment at time of consent, this can be first line platinum based chemotherapy, or immunotherapy, any line.
4. Patients must be ≥ 18 years old.
5. Patients must have provided voluntary written informed consent.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of squamous cell cancer of the head & neck, esophagus, or anal canal who have radiologically confirmed recurrent or metastatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of Genomic, epigenetic and Immune Profiling Features | Through study completion, up to 4 years
  To comprehensively characterize genomic, epigenetic and immune profiling features and changes in longitudinal blood samples that are associated with systemic treatment of recurrent or metastatic squamous cell cancers of the head & neck, esophagus and anal canal.

SECONDARY OUTCOMES:
Establish a Clinically Annotated Biorepository | Through study completion, up to 4 years
  To establish a clinically annotated biorepository of archived tumor and longitudinal blood samples, with serial radiomic evaluations in patients with recurrent/metastatic squamous cell cancers commencing on any new systemic treatments.
Correlate Multi-Omic Results with Clinical Outcome | Through study completion, up to 4 years
  To correlate genomic, othr-omic, radiomic and immune profiling results with clinical outcome - to identify potential predictive markers of response/resistance to systemic therapy.
Compare HPV-Positive and HPV-Negative Cell Histologies | Through study completion, up to 4 years
  To compare HPV-positive and HPV-negative squamous cell histology across three disease sites with multi-omic assessment.
Investigate the Relationship Between Genomic Profiles and Radiomic Signatures | Through study completion, up to 4 years
  To investigate whether any correlation or relation exists between tumor genomic profiles and radiomic imaging signatures.
Enable Data-Sharing | Though study completion, up to 4 years
  To enable data sharing with Queen's University Belfast as a collaborative initiative based on this project

CONTACTS AND LOCATIONS:
Overall Officials: Elena Elimova, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada